CLINICAL TRIAL: NCT00866853
Title: A Phase I, Open Label, 2-period, Randomized, Crossover Trial in 16 Healthy Subjects to Assess the Drug Interaction Potential of TMC435 With Oral Midazolam and With a Drug Cocktail Representative of CYP1A2, CYP2C9, CYP2D6, CYP3A4, and CYP2C19 Substrates.
Brief Title: TMC435-TiDP16-C107: This Study Measures the (Possible) Influence of TMC435 on the Activity of a Selected Set of Drug-degrading Proteins by Measuring the Blood Levels of Drugs That Have Been Taken Together With TMC435 and That Are Known to be Specifically Degraded by These Drug-degrading Proteins.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals Limited, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015949
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C; Viruses
Keywords: TMC435350; HCV; Hepatitis C; TMC435; protease inhibitor; CYP; Cooperstown 5+1 cocktail
MeSH Terms: conditions — Hepatitis C; Virus Diseases | interventions — Simeprevir

INTERVENTIONS:
Drug: TMC435

SUMMARY:
The purpose of this study is to determine whether TMC435 influences the activity of certain drug-degrading proteins in the human body. The drug-degrading proteins investigated in this study belong to the Cytochrome P (CYP) family and are called CYP1A2, CYP2C9, CYP2D6, CYP3A4 and CYP2C19. The activity of these drug-degrading enzymes are determined by measuring the blood levels of a selected set of drugs, which are taken together with TMC435, and, which are known to be specifically degraded by a certain member of the CYP family. This selected set of drugs (which are taken together and therefore called a "drug cocktail") are considered as "probes" of these respective drug-degrading enzymes. By measuring the levels of these probes in human blood, the activity of these degrading enzymes are being revealed. In this way, we can determine if TMC435 influences in one way or another the activity of one or several of these selected drug-degrading proteins.

DETAILED DESCRIPTION:
This is an open-label 2-period randomized cross-over trial in 16 healthy volunteers. Eligible volunteers will be randomized to 2 groups. Volunteers in Group A will receive in Period 1 a single dose of oral midazolam and a drug cocktail alone on Day 1 and 2, respectively (Treatment A). In Period 2, they will receive 150 mg TMC435 once daily on Days 1-11 with a single dose of oral midazolam and a drug cocktail on Day 10 and 11, respectively (Treatment B). Volunteers in Group B will receive in Period 1 Treatment B and in Period 2 Treatment A. There is a period of at least 14 days between the two periods to ensure that all drugs administered in the previous period have been degraded and will not interfere with the measurements of the following period. The cocktail consists of midazolam (administered intravenously (abbreviated as "i.v.", which means directly injected into a blood vein. Injection occurs over a period of 1 minute via a a small tube (canula) that is brought into the blood vein to ease slow injection of the drug), omeprazole, dextromethorphan, caffeine and warfarin. Each of these drugs is being degraded by a specific drug-degrading protein of the CYP family, and are therefore ideal tools to reveal the activity of this specific protein. The amount of TMC435, midazolam, cocktail drugs (and some of their metabolites, i.e. degradation products) in blood will be assessed on selected time points. Safety and tolerability of the coadministration of TMC435 and oral midazolam and of TMC435 and the drug cocktail will be assessed throughout the trial. Safety and tolerability follow up includes the assessment of several blood parameters (blood cells, biochemical activity of certain proteins, minerals, coagulation factors, …), of several parameters in urine (blood cells, proteins, glucose, …) and of the cardiac activity (via electrocardiogram, blood pressure, pulse rate). Healthy volunteers will receive treatments in either A-B sequence or B-A sequence. Treatment A consists of oral midazolam (0.075 mg/kg) on Day1 and cocktail (*) on Day2. Treatment B consists of TMC435 (150 mg q.d.) on Day1-11, oral midazolam (0.075 mg/kg) on Day10 and cocktail (*) on Day11. (*) Cocktail: 0.025 mg/kg midazolam (i.v.), dextromethorphan (30 mg, orally), caffeine (150 mg, orally), omeprazole (40 mg, orally) and warfarin (10 mg, orally) supplemented with vitamin K (10 mg, orally)

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is a non-smoker for at least 3 months prior to screening
* Healthy on the basis of a physical examination, medical history, electrocardiogram, vital signs and the results of blood biochemistry, blood coagulation, and hematology tests and a urinalysis carried out at screening
* Normal weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included

Exclusion Criteria:

* No volunteers who carry certain forms of the CYP2D6, CYP2C9 and CYP2C19 genes, which cause a weak activity of these drug-degrading proteins. These forms are: genotype *3, *4, *5, *6 for CYP2D6, *2, *3 for CYP2C9 or *2, *3, *4, *8 for CYP2C19
* No Hepatitis A, B, or C infection at screening
* No history and/or clinical signs and symptoms of hereditary or acquired coagulation disorders
* No positive Human Immunodeficiency Virus (HIV) 1 or 2 test
* No positive pregnancy test or breast-feeding at screening
* No subjects not using adequate birth control methods.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Plasma levels of TMC435, midazolam and the compounds of the cocktail (+ metabolites) will be assessed. | On defined time points on Day1-6 (Treatment A) and Day1-15 (Treatment B).

SECONDARY OUTCOMES:
To determine the short-term safety and tolerability of the concomitant use of TMC435 and oral midazolam or a cocktail of representative probes of drug-degrading enzymes of the CYP family | On days 1, 2, 3 and 5 of Treatment A and on days 1, 2, 10, 11, 12 and 15 of Tretament B
To determine the steady-state pharmacokinetics of TMC435 given 150 mg once daily | On days 9, 10, 11, 12, 13, 14 and 15 of Treatment B

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited